CLINICAL TRIAL: NCT07182019
Title: Connecting Today to Combat Social Isolation and Loneliness: An Evaluation of a Remote Visiting Program for Care Home Residents Living With Dementia
Brief Title: Connecting Today to Combat Social Isolation and Loneliness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00152323
Record Dates: First submitted 2025-09-16; First posted 2025-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Dementia in Nursing Home; Family; Remote Visits
Keywords: Quality of life; Loneliness; Social support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analyst will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive the Connecting Today intervention for 6 weeks following T0 (i.e. the first outcome data collection period).
  Interventions: Behavioral: Connecting Today
- Control (No Intervention): The control group will not receive the Connecting Today intervention after T0. They are a waitlist control, so will receive the Connecting Today intervention after T1 (i.e. after the second outcome data collection period). Data collection for outcome variables will be the same as participants in the intervention group. The only difference between groups is timing of the intervention.

INTERVENTIONS:
Behavioral: Connecting Today — Connecting today is a facilitated remote visiting program for people living with moderate to severe dementia in care homes. The program offers residents up to 60 minutes of scheduled contact with a family member, friend or volunteer by video call. An onsite facilitator supports the video calls which are delivered via ipad/zoom.
  Arms: Intervention

SUMMARY:
The investigators developed Connecting Today, a feasible and highly acceptable remote visiting program that can support care home residents living with moderate to severe dementia to have video calls with their family members, friends, or care partners. The investigators will recruit 80 residents from 4 care homes, and their family members, friends, or care partners. All participants will be offered 60 minutes of Connecting Today per week for 6 weeks (in either the intervention group, or in the wait-list control group). An onsite care provider will be trained to tailor the video calls, and facilitate positive verbal and non-verbal engagement during the calls. The investigators will evaluate how Connecting Today affects outcomes for residents (quality of life, loneliness, and responsive behaviours) and their remote visitors (quality of life, loneliness, and social support). The investigators will assess how outcomes differ for men, women, and people with different perceptions and experiences of Connecting Today.

DETAILED DESCRIPTION:
Justification For decades, care home residents living with dementia have suffered disproportionately from social isolation (being alone), loneliness (feeling alone), and poor quality of life. Paradoxically, they have also been excluded from intervention research to address these pernicious problems. The investigators developed Connecting Today, a facilitated remote visiting program, to engage care home residents with dementia in positive interactions with their family members, friends, and care partners. Scoping reviews, a mixed methods study, and pilot/ feasibility studies in Alberta support feasibility and high acceptability of Connecting Today.

Purpose This study will evaluate the feasibility of a multi-province RCT of Connecting Today in preparation for a full effectiveness trial.

Objectives

1. Assess feasibility of a pragmatic randomized wait-list control trial of Connecting Today, a remote visiting program, when used in care homes in Alberta, Saskatchewan and Ontario.
2. Examine Connecting Today's hypothesized mechanisms of action within intervention and wait-list control groups.

Research Method/Procedures The investigators will recruit 80 residents living with dementia from 4 total care homes (one each in Alberta, Saskatchewan, and two in Ontario) and their family members, friends, or care partners (1 to 3 for each resident). Participants will receive 6 weeks of Connecting Today: facilitated video calls (up to 60 min weekly). Residents' designated decision-makers will provide consent for resident participation. Research assistants (blinded to assignment status) will collect reliable and valid outcome measures in telephone interviews for residents (via proxy report) and remote visitors (via self-report). Outcomes are measured for all participants at: T0=baseline (weeks 1-2), T1=after 6 weeks of intervention delivery to the treatment group (weeks 9-10), and T2=after 6 weeks of intervention delivery to the control group (weeks 17-18).

The difference between the control group and intervention group is timing of intervention delivery. The intervention group will receive the intervention in weeks 3-8 (i.e. between T0 and T1) and the control group will receive the intervention in weeks 11-16 (i.e. between T1 and T2).

Plan for Data Analysis To address aim 1 (feasibility), the investigators will complete a quantitative assessment of trial and intervention processes including rates of recruitment, retention, attrition, fidelity of intervention delivery, and missing data (compared to pre-specified thresholds), assignment beliefs, treatment experiences and perceptions, and features of usual care.

To address aim 2 (mechanisms of action), the investigators will use generalized estimating equations and a single group before-after design combining intervention and wait-list control groups to complete a within-group outcomes analysis, adjusted for care home cluster and with gender and intervention processes included as covariates/moderators.

ELIGIBILITY:
Inclusion Criteria:

Residents:

* are at least 65 years old
* are diagnosed with any type of dementia
* have a Cognitive Performance Score (CPS) indicating moderate to severe impairment (CPS 3-6).
* to participate, residents must also have people that self identify as a family member or friend of the person with dementia.

Remote visitors:

* are people that self-identify as a family member or friend of the person with dementia
* are people with whom the person with dementia desires contact
* are 18 or older
* understand and speak English.

Exclusion Criteria:

* All remote visitors are required to understand and speak English as this is necessary for the facilitator to support the call and for data to be collected.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Dementia Quality of Life Instrument (DEMQOL- proxy) total score. | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident quality of life will be measured with the Dementia Quality of Life Instrument (DEMQOL- proxy) total score (completed by a family/friend who knows the person living with dementia well). A sum of 31 items (rated on a 4-point scale) generates the total score, where 31 is the worst possible quality of life and 124 is the best possible quality of life. Items relate to how the person living with dementia feels about their daily activities, health and well-being, cognitive functioning, social relationships, and self-concept.
Change in the Dementia Quality of Life - Care Home Instrument (DEMQOL- CH) total score. | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  The Dementia Quality of Life - Care Home instrument (DEMQOL-CH) is a quality of life assessment tool for people living with dementia that is completed by care home staff (i.e. research nurse). There are 31 items rated on a 4-point scale (total score 31-124), where 31 is the worst possible quality of life and 124 is the best possible quality of life.
Change in the the Quality of Life - Aged Care Consumers (QOL-ACC- proxy) total score. | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident quality of life will be measured using the Quality of Life - Aged Care Consumers (QOL-ACC-proxy). It is completed by someone who knows the resident well (in this study both a family/friend proxy and research nurse will complete the measure), and includes questions on health-related and psychosocial aspects of quality of life. There are 6 questions that are answered on a 5 point scale. Total scores range from 0 to 24, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in single item from the Dementia Quality of Life Instrument (DEMQOL- proxy) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident global quality of life will be measured with a single item from the Dementia Quality of Life Instrument (DEMQOL- proxy) completed by a family/friend who knows the person living with dementia well. The single item rates quality of life overall, and is rated on a 4-point scale (total score 1-4), where higher scores indicate higher quality of life.
Change in a single item from the Dementia Quality of Life - Care Home Instrument (DEMQOL- CH) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident global quality of life will be measured with a single item from the Dementia Quality of Life - Care Home Instrument (DEMQOL- CH) completed by care home staff (i.e. research nurse) who knows the person living with dementia well. The single item rates quality of life overall and is rated on a 4-point scale (total score 1-4), where higher scores indicate higher quality of life.
Change in three items from the Dementia Quality of Life Instrument (DEMQOL- proxy) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident loneliness will be measured with three items from the Dementia Quality of Life Instrument (DEMQOL- proxy) (completed by a family/friend who knows the person living with dementia well). These include worries about: (1) getting in touch with people; (2) not having enough company; (3) not being able to help other people. Each item is rated on a 4-point scale (total score 1-4), with higher scores indicating less loneliness. Each will be analyzed as single items.
Change in three items from the Dementia Quality of Life - Care Home Instrument (DEMQOL- CH) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident loneliness will be measured with three items from the Dementia Quality of Life - Care Home Instrument (DEMQOL- CH) completed by care home staff (i.e. research nurse) who knows the person living with dementia well. These include worries about: (1) getting in touch with people; (2) not having enough company; (3) not being able to help other people. Each item is rated on a 4-point scale (total score 1-4), with higher scores indicating less loneliness. Each will be analyzed as single items.
Change in the Social Connection In Long-Term Care Home Residents (SONNET) Scale-proxy | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Change in resident loneliness will be measured by the Social Connection In Long-Term Care Home Residents (SONNET) Scale-proxy, completed by a research nurse. This scale measures overall social connection of residents, as well as their social engagement and social connectedness. There are 12 questions rated on a 4 point scale (total score 0-36), with higher scores indicating higher social connection.
Change in the Cohen-Mansfield Agitation Inventory - short form | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Resident responsive behaviours will be measured using the Cohen-Mansfield Agitation Inventory - short form, and will be completed by a research nurse. This measures the occurrence of 14 resident behaviours in the last 2 weeks (5-point scales). Three factors are calculated (aggressive behavior, physically non-aggressive behavior, and verbally agitated behavior). Scores range from 14 to 70 with higher scores indicating more frequent agitated behaviors.
Change in the 3-item Loneliness Scale total score | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Remote visitor loneliness will be measured using the 3-item Loneliness Scale total score, which is self-reported. Perceptions of companionship are assessed with three items (3-point scale). Scores range from 3 to 9 (higher scores indicate more loneliness).
Change in the Multidimensional Scale of Perceived Social Support (MSPSS) total score | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Remote visitor social support will be measured using the Multidimensional Scale of Perceived Social Support (MSPSS) total score. The MSPSS is comprised of a total of 12 items (on 7 point scales), with 4 items for each subscale (reflecting social support from significant others, family, and friends). The total score is an average, calculated by summing all items (which could range from 12 to 84) and dividing by 12 (higher scores indicate more social support).
Change in the Quality of Life Scale (QOLS) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Remote visitor quality of life will be measured by the Quality of Life Scale (QOLS). This scale includes 16 items (scored on a 7 point scale), with possible scores ranging from 16-112. Higher scores indicate higher quality of life.
Change in the Satisfaction with Life Scale (SWLS) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Remote visitor quality of life will be measured by the Satisfaction with Life Scale (SWLS). This will be self-reported, and includes 5 questions on 7 point scales (total score 5-35). Higher scores indicated higher life satisfaction.
Change in a single item from the World Health Organization Quality of Life (WHOQOL- BREF) | Baseline (T0), after 6 weeks of intervention delivery to the treatment group (T1), and after 6 weeks of intervention delivery to the control group (T2).
  Remote visitor quality of life will be measured by a single item from the World Health Organization Quality of Life (WHOQOL- BREF). This will be self-reported, and includes responding on a 5 point scale (total score 1-5). The higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah O'Rourke, PhD, Principal Investigator — University of Alberta; Matthias Hoben, Dr rer medic, Principal Investigator — York University; Shelley Peacock, PhD, Principal Investigator — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: No